CLINICAL TRIAL: NCT04447820
Title: A Multicenter, Randomized, Open-Label, 4-Week Study to Investigate the Efficacy and Pharmacokinetic Profile of K-877-ER Once Daily Treatment Compared to K-877-IR Twice Daily Treatment in Adult Patients With Fasting Triglyceride Levels
Brief Title: Study to Investigate the Efficacy and Pharmacokinetic Profile of K-877-ER Compared to K-877-IR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K-877-ER-201
Record Dates: First submitted 2020-06-19; First posted 2020-06-25 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-11

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- K-877-ER Dose A (Experimental): K-877-ER dose A administered once daily
  Interventions: Drug: K-877-ER (Dose A)
- K-877-ER Dose B (Experimental): K-877-ER dose B administered once daily
  Interventions: Drug: K-877-ER (Dose B)
- K-877-IR (Experimental): K-877-IR administered twice daily.
  Interventions: Drug: K-877-IR

INTERVENTIONS:
Drug: K-877-ER (Dose A) — Dose A Oral Administration
  Arms: K-877-ER Dose A
Drug: K-877-ER (Dose B) — Dose B Oral Administration
  Arms: K-877-ER Dose B
Drug: K-877-IR — K-877-IR Oral Administration
  Arms: K-877-IR

SUMMARY:
A study to evaluate the efficacy of K-877 extended release (ER) once daily (QD) compared to K-877 immediate release (IR) twice daily (BID).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent before any study-specific evaluation is performed
* At screening, have a mean fasting TG level of ≥180 mg/dL and <550 mg/dL; at subsequent Qualification Period visits confirm fasting TG level of ≥200 mg/dL and <500 mg/dL
* Able to meet all inclusion criteria outlined in clinical study protocol

Exclusion Criteria:

* Require lipid-altering treatments other than study drugs, statins, ezetimibe, or PCSK9 inhibitors during the study
* Known hypersensitivity or intolerance to fibrates or peroxisome proliferator-activated receptor alpha agonists
* Meet any other exclusion criteria outlined in clinical study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-06-10 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Pinnacle Research Group, Anniston, Alabama
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Columbus Regional Health, Columbus, Georgia
  - Prism Research, Saint Paul, Minnesota
  - Diabetes and Endocrinology Consultants, P.C., Morehead City, North Carolina
  - Medpace Clinical Pharmacology, LLC, Cincinnati, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Summit Research Group, LLC, Munroe Falls, Ohio
  - Health Concepts, Rapid City, South Dakota
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Manassas Clinical Research Center, Manassas, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Screening Period occurred no more than 70 days and no less than 7 days prior to the first dose of study drug. The up to 10-week Screening Period allowed for a 6-week washout period, if needed, followed by an up to 4-week Qualification Period that was used to assess patient eligibility. Prior to treatment on Day 1, eligible patients were randomized in a 1:1:1 ratio to 1 of 3 treatment groups. Randomization was stratified by sex, statin use, and PK assessment.
Groups:
- K-877-IR: K-877 Immediate release (IR) tablet orally twice daily (BID) from day 1 through 28.
- K-877-ER Dose A: K-877 Extended release (ER) tablet (Dose A) orally once daily (QD) from day 1 through 28.
- K-877-ER Dose B: K-877 Extended release (ER) tablets (Dose B) orally once daily (QD) from day 1 through 28.
Period: Overall Study
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
Started | 32 | 32 | 32
Completed | 31 | 31 | 29
Not Completed | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was defined as all randomized patients who took at least 1 dose of study drug and had a baseline fasting TG assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B | Total
Number analyzed (Participants) | 32 | 32 | 32 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 24 | 26 | 22 | 72
  >=65 years | 8 | 6 | 10 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 14 | 44
  Male | 17 | 17 | 18 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 7 | 22
  Not Hispanic or Latino | 24 | 23 | 25 | 72
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 31 | 31 | 31 | 93
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Statin Use [Count of Participants; unit: Participants]
  Yes | 15 | 15 | 15 | 45
  No | 17 | 17 | 17 | 51
TG at Baseline [Mean (Standard Deviation); unit: mg/dL] | 278.72 (53.316) | 294.88 (61.949) | 307.35 (73.575) | 293.65 (63.915)

OUTCOME MEASURES:

1. Primary Outcome: Estimated Percentage Change in Fasting Triglyceride(s) (TG)
Time Frame: Baseline to Day 28
Population: The Per-Protocol Set (PPS) was defined as all patients in the Full Analysis Set without any major protocol deviations and who had baseline and Day 28 fasting serum TG measurements.
Measure: Least Squares Mean (Standard Deviation); unit: Percent Change
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
Number analyzed (Participants) | 31 | 30 | 27
Percent Change | -41.57 (3.295) | -36.79 (3.319) | -38.94 (3.553)
Statistical Analysis 1: Comparison: K-877-IR vs K-877-ER Dose A; Test type: Non-Inferiority — Approximately 90 participants were planned. Assuming an effect size delta = 0, pooled SD = 21.38, an alpha = 0.05 (1-sided), and a non-inferiority limit of 15%, a sample size of 26 patients per treatment group provided a power of 0.80. In the case that the actual effect size delta was 10%, the power was then 0.2. If the real effect was different, the result less likely showed non-inferiority. To account for any potential drop off, 30 participants in each treatment group, were planned; p = 0.3084, Mixed Model for repeated measures (MMRM)
Statistical Analysis 2: Comparison: K-877-IR vs K-877-ER Dose B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.5930, Mixed Model for repeated measures (MMRM)

2. Secondary Outcome: Percentage Change From Baseline to Day 28 in Total Cholesterol (TC)
Time Frame: Baseline to Day 28
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
Number analyzed (Participants) | 31 | 30 | 27
Percent Change | -6.07 (15.417) | -8.68 (13.266) | 0.28 (18.100)
Statistical Analysis 1: Comparison: K-877-IR vs K-877-ER Dose A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.9788, MMRM
Statistical Analysis 2: Comparison: K-877-IR vs K-877-ER Dose B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1314, MMRM

3. Secondary Outcome: Percentage Change From Baseline to Day 28 in Low-density Lipoprotein Cholesterol (LDL-C)
Time Frame: Baseline to Day 28
Population: PPS
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
Number analyzed (Participants) | 31 | 30 | 27
Percent Change | 3.56 (28.586) | -2.16 (21.394) | 22.71 (64.420)
Statistical Analysis 1: Comparison: K-877-IR vs K-877-ER Dose A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.8840, MMRM analysis
Statistical Analysis 2: Comparison: K-877-IR vs K-877-ER Dose B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.1202, MMRM analysis

4. Secondary Outcome: Percentage Change From Baseline to Day 28 in High-density Lipoprotein Cholesterol (HDL-C)
Time Frame: Baseline to Day 28
Population: PPS
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
Number analyzed (Participants) | 31 | 30 | 27
Percent Change | 12.22 (27.335) | 15.39 (18.190) | 20.04 (24.370)
Statistical Analysis 1: Comparison: K-877-IR vs K-877-ER Dose A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.9353, MMRM
Statistical Analysis 2: Comparison: K-877-IR vs K-877-ER Dose B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3099, MMRM

5. Secondary Outcome: Percentage Change From Baseline to Day 28 in Remnant Cholesterol
Time Frame: Baseline to Day 28
Population: PPS
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
Number analyzed (Participants) | 31 | 30 | 27
Percentage Change | -33.85 (32.467) | -30.08 (25.394) | -32.34 (24.761)
Statistical Analysis 1: Comparison: K-877-IR vs K-877-ER Dose A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.2098, MMRM
Statistical Analysis 2: Comparison: K-877-IR vs K-877-ER Dose B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3688, MMRM

6. Secondary Outcome: Percentage Change From Baseline to Day 28 in Non-HDL-C
Time Frame: Baseline to Day 28
Population: PPS
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
Number analyzed (Participants) | 31 | 30 | 27
Percent Change | -10.04 (21.704) | -11.12 (18.847) | -3.74 (21.394)
Statistical Analysis 1: Comparison: K-877-IR vs K-877-ER Dose A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.5647, MMRM
Statistical Analysis 2: Comparison: K-877-IR vs K-877-ER Dose B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.2170, MMRM

7. Secondary Outcome: Percentage Change From Baseline to Day 28 in Free Fatty Acid (FFAs)
Time Frame: Baseline to Day 28
Population: PPS
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
Number analyzed (Participants) | 31 | 30 | 27
Percent Change | -7.35 (45.110) | -17.17 (25.430) | -10.22 (40.436)
Statistical Analysis 1: Comparison: K-877-IR vs K-877-ER Dose A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.2562, MMRM
Statistical Analysis 2: Comparison: K-877-IR vs K-877-ER Dose B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.4268, MMRM

8. Secondary Outcome: K-877 PK Parameters Cmax
Description: Observed maximum measured plasma concentration (Cmax)
Time Frame: Day 28
Population: The PK Analysis Set included all patients from the Safety Analysis Set who had at least 1 PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
Number analyzed (Participants) | 6 | 8 | 7
ng/mL | 2.061 (63.9) | 2.746 (85.2) | 5.433 (61.2)

9. Secondary Outcome: K-877 PK Parameters AUC (Tau)
Time Frame: Day 28
Population: The PK Analysis Set included all patients from the Safety Analysis Set who had at least 1 PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h-ng/mL
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
Number analyzed (Participants) | 5 | 8 | 7
h-ng/mL | 10.239 (43.1) | 22.566 (71.3) | 41.611 (44.1)

ADVERSE EVENTS:
Time Frame: 28 Days
Description: 1. The Safety Analysis Set was defined as all randomized participants who received at least 1 dose of the randomized study drug.
  2. Treatment-emergent AEs (TEAEs) were defined as AEs that occurred for the first time after the first dose of study drug or existed prior to the first dose and worsened during the Treatment Period.
Arm/Group | K-877-IR | K-877-ER Dose A | K-877-ER Dose B
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 1/32 | 5/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | K-877-IR (N=32) | K-877-ER Dose A (N=32) | K-877-ER Dose B (N=32)
Headache (Nervous system disorders) | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol: Ver: 1.0 (2020-01-28): https://cdn.clinicaltrials.gov/large-docs/20/NCT04447820/Prot_000.pdf
  • Study Protocol: Ver: 2.0 (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/20/NCT04447820/Prot_001.pdf
  • Statistical Analysis Plan: Ver 1.0 (2020-08-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT04447820/SAP_002.pdf
  • Statistical Analysis Plan: Ver 2.0 (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT04447820/SAP_003.pdf